CLINICAL TRIAL: NCT04378049
Title: Robot-Assisted Partial Knee Replacement Versus Standard Total Knee Replacement: A Pilot Randomized Controlled Trial
Brief Title: Robot-Assisted Partial Knee Replacement Versus Standard Total Knee Replacement
Acronym: RoboKnees
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Hamilton Academic Health Sciences Organization (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RoboKnees
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; Unicompartmental knee arthroplasty; Robot-assisted surgery; Pilot randomized controlled trial; Bicompartmental knee arthroplasty; Mako partial knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Masking Description: Surgeons cannot be blinded to treatment group. It would not be feasible to blind the health care team and patients because the incisions and imaging are visually distinguishable. We will attempt to minimize bias in subjective measures by presenting patients with balanced information on each treatment group prior to the trial. All participants will receive a computed tomography (CT) scan prior to surgery to maintain blinding and to give surgeons additional information about 3 dimensional modelling for implant placement. Data analysts will be blinded to treatment allocation. An independent outcomes assessor will independently review radiographic alignment for each patient and review relatedness of adverse events and re-operations. The independent assessor cannot be blinded because imaging is visually distinguishable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard total knee arthroplasty (Active Comparator): Participants who are randomized to the control group will undergo TKA according to local standard of care. The choice of implant and use of bone cement will be recorded but left to the surgeon's discretion according to their standard practice.
  Interventions: Procedure: Total knee arthroplasty
- Robot-assisted partial knee arthroplasty (Experimental): Participants with isolated medial or isolated lateral compartment OA who are randomized to the intervention group and have one affected knee compartment will receive a robot-assisted unicompartmental knee arthroplasty (UKA). If the patient has medial or lateral OA plus patellofemoral OA they will receive a bicompartmental knee arthroplasty (BiKA) consisting of a two simultaneous UKAs. The partial knee replacement procedures will be performed using the Mako RIO robotic arm (Stryker) according to the manufacturer's instructions. The choice of implant and use of bone cement will be recorded but will be left to the surgeon's discretion. Surgeons will resurface the patella if the patellar cartilage meets Outerbridge grade 3 or 4 criteria
  Interventions: Procedure: Robot-assisted partial knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Surgeon will perform a total knee arthroplasty procedure according to local standard of care
  Other Names: Total knee replacement
  Arms: Standard total knee arthroplasty
Procedure: Robot-assisted partial knee arthroplasty — Surgeon will perform a robot-assisted unicompartmental or bicompartmental knee arthroplasty procedure
  Other Names: MakoPlasty
  Arms: Robot-assisted partial knee arthroplasty

SUMMARY:
This is a pilot randomized trial to assess the feasibility of a definitive trial to determine the effect of robot-assisted partial knee replacements versus standard total knee replacements.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) pain is an important source of morbidity and cost to the health care system. Over 60,000 knee replacement surgeries are performed in Canada every year, making it the second most common surgery. Our institution (St. Joseph's Healthcare Hamilton) is the first hospital in Canada to purchase a Mako RIO orthopaedic robot to assist with performing knee replacements. The knee is divided into three compartments, and one, two, or all three compartments can become arthritic. Over 90% of patients with end-stage knee OA receive a total knee replacement (also known as total knee arthroplasty or TKA) even if they have one or two healthy knee compartments. Partial knee replacements are an option for these patients but these procedures are very technically demanding and associated with a higher risk of implant failure. For this reason, few surgeons are experts at partial knee replacements. We believe that we can use robotic technology to make it easier for surgeons to perform partial replacements more accurately, thereby increasing the quality and survivorship of partial knee replacements. This may lead to better patient-important outcomes like return to activity, pain, and satisfaction, and eventually better access to high-quality partial knee replacements for Canadians. This will be the first study to evaluate total knee replacements (standard care) versus robot-assisted partial knee replacements, and could lead to greater uptake of robotic technology in orthopaedics and a shift toward anatomy-sparing partial knee replacements.

ELIGIBILITY:
Inclusion criteria

* Adult (18+)
* Unicompartmental knee OA with or without concomitant patellofemoral OA, requiring surgical treatment
* Two study surgeons independently agree that the patient is eligible for either treatment group

Exclusion criteria

* Inability to provide informed consent (e.g. cognitive disability, language barrier)
* Revision knee surgery
* Simultaneous bilateral knee surgery
* Previous major knee surgery or trauma
* The robot or required components are unavailable (e.g. technical difficulties, robot-specific disposables out of stock)
* A CT scan cannot be obtained prior to surgery
* Patient does not wish to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility- Recruitment | 12 months
  The number of patients recruited during a 12 month period
Feasibility- Participant retention | 12 months
  Number of patients completing the study
Feasibility- Treatment compliance | 12 months
  The number of crossovers during a 12 month period

SECONDARY OUTCOMES:
Return to function questionnaire | 12 months post-surgery
  We will use the 5-item Return To Function (RTF) questionnaire to determine when a trial participant returns to work, leisure, and activities around the home after an injury or surgery (measured as time to return to unrestricted activities).
Oxford knee score | 12 months post-surgery
  We will measure knee function using the Oxford Knee Score (OKS), which is a validated and well-used 12 item questionnaire used to measure knee function when performing daily activities after total knee replacement surgery. The OKS is scored on a 0-48 scale with higher scores representing a better outcome.
Forgotten joint score | 12 months post-surgery
  We will use the Forgotten Joint Score (FJS-Knee) to measure how natural the replaced knee feels. The FJS-Knee is a 12 item questionnaire that aims to assess both function and feeling by asking about patients' awareness of their artificial knee while doing various daily activities. The FJS is scored on a 0-100 scale with higher scores representing a better outcome.
Gait walking mechanics analysis | 12 months post-surgery
  Overground walking kinematic gait analysis will be performed in the clinic environment using a ten-camera optoelectronic motion capture system. Primary gait outcomes will include the knee joint flexion and adduction angle magnitudes and range during the stance phase of gait. Secondary gait outcomes will include stride characteristics as defined above, knee transverse rotation during stance, knee flexion during swing, hip and ankle range of motion and peak magnitudes during stance.
Quality of life- EQ-5D | 12 months post-surgery
  We will use the Euro-Qol 5 Dimensions (EQ-5D) questionnaire, a widely used and well-validated quality of life tool, to measure participant quality of life. The EQ-5D is a comprehensive, 5-item compact health status classification and health state preference questionnaire.
Persistent post-surgical pain (PPSP) | 12 months post-surgery
  We will use a modified version of the WHO's definition of PPSP, to include a minimum threshold of pain severity:
  1. Pain that began after surgery or a tissue trauma;
  2. Pain is in an area of preceding surgery or tissue trauma;
  3. Pain has persisted for at least three months after surgery; and
  4. The pain is not better explained by an infection, malignancy, a pre-existing pain condition or any other alternative cause.
  5. ≥4 out of 10 on the numeric rating scale (NRS) from the Brief Pain Inventory (BPI-SF) for "average pain over the last week". The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine)
Patient global impression of change score | 12 months post-surgery
  We will use The Patient Global Impression of Change (PGIC) scale to assess patients' beliefs about the efficacy of treatment. The PGIC is one item and asks patients to rate the effectiveness of the treatment of interest on a 7-point ordinal scale ranging from "very much improved" to "very much worse
Healthcare resource use (for cost-effectiveness) | 12 months post-surgery
  We will collect healthcare resource utilization information (e.g. hospitalization, physician visits) and information on productivity (e.g. time missed from work) to assist with health economic analyses.
Rage of motion (ROM) | 6 weeks post-surgery
  We will measure knee ROM using a goniometer at in-clinic visits according to standard practice
Knee alignment | Post-surgery
  We will measure mechanical alignment on pre-operative and post-operative weightbearing x-rays
Adverse events | 12 months post-surgery
  We will collect all serious adverse events and surgery-related non-serious adverse events throughout the trial for safety monitoring purposes
Short-term implant survival | 12 months post-surgery
  We will report the number of revision surgeries within the study period including cases of periprosthetic joint infection, aseptic loosening, instability, poly wear, intractable pain, periprosthetic fracture etc.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Adili, MD, P.Eng, FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will share data upon reasonable request for non-commercial purposes. This may require an institutional data-sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon study completion.

REFERENCES:
- [Derived] Madden K, Flood B, Malek M, Milantoni V, Astephen Wilson JL, Tarride JE, Khanna V, Adili A; RoboKnees Investigators. Robot-assisted partial knee replacement versus standard total knee replacement (RoboKnees): a protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2024 Feb 21;10(1):39. doi: 10.1186/s40814-024-01463-x. PMID 38383530